CLINICAL TRIAL: NCT06745492
Title: Low-dose Neostigmine at TOF Ratio of 0.7 Accelerates Neuromuscular Recovery Without Adverse Effects: a Prospective Observational Study
Brief Title: Low-dose Neostigmine at TOF Ratio of 0.7 Improves Neuromuscular Recovery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang-Hoon Koo, Professor, Seoul National University Bundang Hospital
Other Study IDs: Neostigmine & TOFR 0.7
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Recovery Time
MeSH Terms: interventions — Neostigmine; Glycopyrrolate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Neostigmine + Glycopyrrolate — a 20 mcg/kg of neostigmine and 4 mcg/kg of glycopyrrolate were administered at a TOF ratio of 0.7.

SUMMARY:
This study is a prospective observational study. A total of 54 patients were included in this study. We observed the time from neostigmine administration to TOF ratio of 1.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective thyroid surgery under general anesthesia
* a body mass index of 18.5-25 kg/m2
* Age ≥ 20

Exclusion Criteria:

* Refused to participate
* history of hypersensitivity to acetylcholinesterase inhibitor
* neuromuscular disease
* hepatic or renal dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective thyroid surgery under general anesthesia were screened and included in this study
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Recovery time | During surgery
  Time from neostigmine administration to TOF ratio of 1.0

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hoon Koo, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No